CLINICAL TRIAL: NCT01419678
Title: Pharmacokinetic Analysis of Posaconazole in Lung Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO10110232
Record Dates: First submitted 2011-08-12; First posted 2011-08-18 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Lung Transplant Infection; Fungal Infection
Keywords: posaconazole; PK blood sampling
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 'collection of blood samples for PK testing' (Experimental): collection of PK samples around a dosing of Posaconazole
  Interventions: Other: collection of blood samples for PK testing

INTERVENTIONS:
Other: collection of blood samples for PK testing — PK samples collected around dosing of posaconazole

SUMMARY:
This is a single center, observational study of posaconazole PK sampling in lung transplant recipients. The patients enrolled will have up to 6 (3ml) pk samples (a total of 18 ml) and one 10ml blood sample for a total collection of 28ml of blood obtained over the entire study. In addition, the investigators will collect medical record information and any excess BAL samples available during the study (tests done as part of the patient's clinical care and the samples would have been discarded once diagnosis was made).

DETAILED DESCRIPTION:
PK blood samples will be obtained around a clinical dosing of posaconazole

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older receiving posaconazole post transplant as part of their care received a lung transplant

Exclusion Criteria:

* must meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
measure the levels of posaconazole post dosing | 24 hours after dosing
  pk samples will be obtained around dosing of medication and then analyzed for posaconazole levels

SECONDARY OUTCOMES:
determine the posaconazole concentration within the pulmonary epithelial lining fluid (ELF) and alveolar cells | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Shields, Pharm D, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States